CLINICAL TRIAL: NCT02575079
Title: Parafilm Application to Prevent Central Line Associated Bloodstream Infections in Pediatric Patients Undergoing Hematopoietic Cell Transplantation
Brief Title: Parafilm to Prevent CLABSI in Pediatric Patients Undergoing HCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Lakshmanan Krishnamurti, Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00080344
Record Dates: First submitted 2015-10-12; First posted 2015-10-14 (Estimated); Results first posted 2019-06-25 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Central Line Associated Bloodstream Infections (CLABSI); Bone Marrow Transplant

STUDY DESIGN:
Intervention Model Description: Arm 1 is comprised of study participants receiving parafilm applied over the CVC hub or around the CVC hub connection. Arm 2 is a retrospective historical cohort of pediatric patients receiving HCT for the purpose of comparing CLABSI rates.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Parafilm (Experimental): Pediatric patients undergoing hematopoietic stem cell transplant (HCT) with central venous catheters (CVCs) will have pre-cut, single-use sections of parafilm applied over the CVC hub (if not connected) or around the CVC hub connection (if connected). Parafilm will be maintained on the CVC and routine CVC care will be continued, per institutional standard of practice, until the CVC is removed.
  Interventions: Device: Parafilm
- Historical Cohort (No Intervention): Pediatric patients receiving hematopoietic cell transplantation in the 16 months preceding the study intervention. Data were obtained retrospectively through medical records for the purpose of comparing CLABSI rates among recipients of parafilm to a control group.

INTERVENTIONS:
Device: Parafilm — Single-use, pre-cut sections of parafilm over the central venous catheter (CVC) hub (if not connected) or around the CVC hub connection (if connected). Parafilm will be maintained on the CVC until it is removed.
  Arms: Parafilm

SUMMARY:
The purpose of this study is to see if applying parafilm as an external barrier on the central line in children having a bone marrow transplant helps to prevent central line associated bloodstream infection(s) and also to assess the ease of use of parafilm.

DETAILED DESCRIPTION:
Central line associated bloodstream infections (CLABSI) result in significant morbidity and mortality, particularly in patients undergoing hematopoietic cell transplantation (HCT). HCT patients are at high risk for CLABSI due to multiple factors, including prolonged immune suppression and the need for long-term central venous access. The investigators want to assess the feasibility of the use of a parafilm central line barrier (parafilm) as standard of care in pediatric HCT patients. The investigators will also assess the effectiveness of the parafilm to reduce the incidence of CLABSI in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Must be between the age of 0 and 21 years at the time of enrollment
* Must be undergoing allogeneic or autologous HCT for a malignant or non-malignant disorder
* Must have or be scheduled to have a tunneled CVC

Exclusion Criteria:

* Patients undergoing other interventions to prevent CLABSI (e.g. Children's Oncology Group (COG) study ACCL1034 with Chlorhexidine Gluconate (CHG); antimicrobial lock therapy, etc.)
* Patients who only have a port

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 119 (Actual)
Dates: Start 2015-03; Primary Completion 2018-03-29 (Actual); Study Completion 2018-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lakshmanan Krishnamurti, MD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States

REFERENCES:
- [Result] Stenger EO, Newton JG, Leong T, Kendrick L, McManus L, Rooke C, Krishnamurti L. Application of parafilm as a physical barrier on CVC connections is feasible and may reduce CLABSI among pediatric HCT patients. Biology of Blood Marrow Transplantation 25 (Suppl 3): S131, 2019.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in the parafilm study between March 2015 and June 2017. All study procedures and follow up was completed on March 29, 2018.
Pre-assignment Details: Fifty-one individuals consented to participate in the study. Prior to beginning any study interventions one was lost to follow up, one withdrew, and one did not begin the prep regimen, resulting in 48 participants who began the study intervention.
Groups:
- Parafilm: Pediatric patients undergoing hematopoietic stem cell transplant (HCT) with central venous catheters (CVCs) who had pre-cut, single-use sections of parafilm applied over the CVC hub (if not connected) or around the CVC hub connection (if connected).
Period: Overall Study
Arm/Group | Parafilm | Historical Cohort
Started | 48 | 71
Completed | 42 | 71
Not Completed | 6 | 0
Not completed — Death | 3 | 0
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Parafilm | Historical Cohort | Total
Number analyzed (Participants) | 48 | 71 | 119
Age, Customized [Count of Participants; unit: Participants]
  Age in years: Less than or equal to 2 years | 7 | 21 | 28
  Age in years: Between 3 and 9 years | 25 | 22 | 47
  Age in years: Between 10 and 21 years | 16 | 28 | 44
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 25 | 42
  Male | 31 | 46 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 6 | 14
  Not Hispanic or Latino | 40 | 65 | 105
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Asian | 0 | 4 | 4
  Ethnicity: Black or African American | 21 | 32 | 53
  Ethnicity: White | 25 | 34 | 59
  Ethnicity: Other | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 48 | 71 | 119
Type of HCT [Count of Participants; unit: Participants]
  Allogeneic | 35 | 49 | 84
  Autologous | 13 | 22 | 35
Underlying disease [Count of Participants; unit: Participants]
  Malignant, hematologic | 17 | 24 | 41
  Malignant, solid tumor | 12 | 21 | 33
  Non-malignant | 19 | 26 | 45

OUTCOME MEASURES:

1. Primary Outcome: Rate of Central Line Associated Bloodstream Infections (CLABSI)
Description: Central line associated bloodstream infections (CLABSI) is the identification of a bacterial infection from a blood culture drawn from a central venous catheter (CVC) in the absence of a primary source of infection from another body site. The CLABSI rate (total number of CLABSI/1000 catheter-days) in parafilm study participants will be calculated and compared to the CLABSI rate in a historical cohort of pediatric patients who are serving as a control group.
Time Frame: Baseline (at the time of placement of the CVC or admission for HCT, whichever occurs later) to end of study (CVC removal or transfer back to primary service, whichever occurs sooner, average of 3 months)
Measure: Number (95% Confidence Interval); unit: CLABSI/1000 catheter-days
Arm/Group | Parafilm | Historical Cohort
Number analyzed (Participants) | 48 | 71
CLABSI/1000 catheter-days | 3.69 [2.19 to 5.83] | 4.37 [2.86 to 6.40]

2. Primary Outcome: Reported Inpatient Percentage of Central-line Days With Correctly Applied Parafilm
Description: In the inpatient setting, compliance was measured by once daily recording of parafilm change by nursing in the electronic medical record. These data were significantly limited by electronic medical record charting on parafilm change being required only once per day. Thus, once daily data collection failed to capture daily parafilm change, given multiple nursing shifts on a single calendar day. Nonetheless, the percentage of catheter-days with intact correctly applied parafilm, as reported by nursing staff, was calculated.
Time Frame: At discharge (an expected average of 6 weeks from admission)
Population: Participants in the parafilm study are included in this analysis. Percentage of inpatient days where nursing charted parafilm change in the electronic medical record is reported for the entire parafilm cohort.
Measure: Number; unit: percentage of central-line days
Arm/Group | Parafilm
Number analyzed (Participants) | 48
percentage of central-line days | 65.2

3. Primary Outcome: Observed Inpatient Percentage of Catheter-days With Correctly Applied Parafilm
Description: Observed compliance occurred during weekly line rounds. Rounding providers indicated whether a patient's parafilm is intact and correctly applied, not applied, or incorrectly applied or not intact. The percentage of "observed catheter-days" where patients had correct use of intact parafilm were to be calculated. To track observed inpatient compliance with applying parafilm, data fields were added to the entered to the nursing charts of the participant's electronic medical record (EMR). The primary field added was a no/question about parafilm applied. Per study protocol, the intent was to document nursing changing of the parafilm, at the time it was changed. However, on reviewing the data, it appears that nursing just charted once per day whether they had changed parafilm or not, while the parafilm may have been changed earlier by a different nurse.
Time Frame: Time between initial bone marrow transplant (BMT) discharge and either central venous line (CVL) removal or transfer back to primary MD (an expected average of 2-3 months)
Population: The data collected indicated that nursing staff did not understand how the parafilm monitoring needed to be charted for the purposes of data analysis. Although a data field was created in the EMR, in practice, the data collected was not an accurate assessment of parafilm use, thus no data are available for analysis of this outcome measure.
Arm/Group | Parafilm
Number analyzed (Participants) | 0

4. Primary Outcome: Reported Outpatient Percentage of Catheter-days With Correctly Applied Parafilm
Description: For outpatient reported compliance, parents of study participants provided their logs to outpatient staff who documented the number of days parafilm was correctly in use/intact vs not in use or incorrectly in use/not intact. The cumulative percentage of catheter-days where parafilm was intact was calculated.
Time Frame: as for outcome 1
Population: The population used for this analysis consists of caretakers who returned outpatient logs of parafilm use at the end of the study. Forty-one participants used parafilm in the outpatient setting and of these 34 returned the outpatient logs.
Measure: Number; unit: percent of catheter-days
Arm/Group | Parafilm
Number analyzed (Participants) | 34
percent of catheter-days | 64.7

5. Primary Outcome: Observed Outpatient Percentage of Catheter-days With Correctly Applied Parafilm
Description: For observed compliance, the outpatient nurse recorded whether the patient's parafilm was correctly applied/intact (yes), not applied (no), or incorrectly applied/not intact (yes-inc) at the beginning of the visit. The percentage of outpatient "observed catheter-days" where parafilm was correctly in use/intact was calculated.
Time Frame: Time between initial BMT discharge and either CVL removal or transfer back to primary MD (an expected average of 2-3 months)
Population: Observed outpatient compliance was not performed as it was difficult to implement this in a busy clinic setting.
Arm/Group | Parafilm
Number analyzed (Participants) | 0

6. Secondary Outcome: Number of Antibiotic Treatment Courses Per Participant
Description: The number of antibiotic treatment courses per participant in the parafilm study will be recorded.
Time Frame: as for outcome 1
Population: Data on antibiotic treatment courses were not collected.
Arm/Group | Parafilm
Number analyzed (Participants) | 0

7. Secondary Outcome: Duration of Antibiotic Treatment Exposure
Description: Total duration of antibiotic treatment exposure (excluding prophylactic antibiotics) among participants in the parafilm study will be reported.
Time Frame: as for outcome 1
Population: Data on duration of antibiotic treatments were not collected.
Arm/Group | Parafilm
Number analyzed (Participants) | 0

8. Secondary Outcome: Number of ICU Admissions Secondary to Sepsis
Description: The cumulative number of ICU admissions secondary to sepsis among participants in the parafilm study is reported.
Time Frame: as for outcome 1
Population: Participants in the parafilm study are included in this analysis.
Measure: Number; unit: ICU admissions
Arm/Group | Parafilm
Number analyzed (Participants) | 48
ICU admissions | 8

9. Secondary Outcome: Death
Description: Deaths from infection and death from any cause among participants in the parafilm study are reported.
Time Frame: as for outcome 1
Population: Participants in the parafilm study are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Parafilm
Number analyzed (Participants) | 48
Participants
  Death from infection | 0
  Death from any cause | 3

10. Secondary Outcome: Perception of Parafilm
Description: The perception of parafilm from provider and caregiver surveys regarding parafilm ease of use, perceived benefit, and other parameters will be reported
Time Frame: Month 3 (average time till removal of CVC)
Population: A survey was initially planned for in the protocol but was removed from the study procedures prior to any participants completing the survey.
Arm/Group | Parafilm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time a participant entered the study until CVC removal (3 months on average).
Description: Adverse events will be described using event terms and severity grading from the National Cancer Institute (NCI) CTCAE version 4.0. Adverse events will be characterized by severity grading, attribution (relationship to study treatment), and expectedness (based upon prior experience). Only unexpected serious adverse events and serious adverse events related to the study intervention were collected. Non-serious adverse events were not collected.
Arm/Group | Parafilm
All-Cause Mortality (participants affected / at risk) | 3/48
Serious Adverse Events (participants affected / at risk) | 3/48
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Parafilm (N=48)
Acute hypoxemic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Graft versus host disease (GVHD) (Immune system disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Assessing feasibility of outpatient parafilm use was limited by difficulty collecting parafilm compliance calendars from caretakers and observed variability of compliance in the outpatient setting.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-24): https://cdn.clinicaltrials.gov/large-docs/79/NCT02575079/Prot_SAP_000.pdf